CLINICAL TRIAL: NCT03657082
Title: Effects of Positive Expiratory Pressure on Inspiratory Capacity and Dyspnea in Patients With COPD During Exercise
Brief Title: Effects of PEP on IC During IT in Patients With COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No financial support found
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, William Poncin, PT, PhD, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PEP-IC
Record Dates: First submitted 2018-08-28; First posted 2018-09-04 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): In this arm, patients will receive the experimental condition first, then the sham condition
  Interventions: Device: PEP-10; Device: PEP-1
- Arm B (Experimental): In this arm, patients will receive the sham condition first, then the experimental condition
  Interventions: Device: PEP-10; Device: PEP-1

INTERVENTIONS:
Device: PEP-10 — Bottle PEP with a water level of 10 cmH2O
Device: PEP-1 — Bottle PEP with a water level of 1 cmH2O

SUMMARY:
This study will investigate the effects of positive expiratory pressure (PEP) on hyperinflation in patients with chronic obstructive pulmonary disease (COPD). Inspiratory capacity (IC) is the primary outcome

DETAILED DESCRIPTION:
This is a cross-over intervention assessing the effect of PEP on IC and dyspnea in patients with COPD performing an interval training (IT) session.

IC will be measured before, during and immediately after the IT session. Each participant will receive perform IT sessions including either the use of a PEP of 10 cmH2O or a PEP of 1 cmH2O. The effects on IC and dyspnea on both PEP levels will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Stable COPD since 1 month at least
* Able to understand the instructions

Exclusion Criteria:

* COPD with a forced expiratory volume at one second > 80% of predicted values
* In exacerbation
* Orthopedic of neurological condition likely to interfere with the experimentation
* Contraindication to perform exercise

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change in inspiratory capacity | 20 minutes
  Evolution of inspiratory capacity while performing the interval training session

SECONDARY OUTCOMES:
Change in Borg scale | 20 minutes
  Evolution of dyspnea while performing the interval training session

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium